CLINICAL TRIAL: NCT04339257
Title: Which Patients With a ROSC After OHCA Would Potentially Benefit From Physician Driven Post Cardiac Arrest Care?
Brief Title: Pre-hospital Post ROSC Care: Are we Achieving Our Targets?
Acronym: POP-ROC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Fabian Lucassen, Principal Investigator, University Medical Center Groningen
Other Study IDs: 201900756
Record Dates: First submitted 2020-03-16; First posted 2020-04-09 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Post Cardiac Arrest Syndrome; Emergency Medical Services
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rational: Out of hospital cardiac arrest is a devastating event with a high mortality. Survival rates have increased over the last years, with the availability of AED's and public BLS. Previous studies have shown that deranged physiology after return of spontaneous circulation (ROSC) is associated with a worse neurological outcome. Good quality post-arrest care is therefore of utmost importance.

Objective: To determine how often prehospital crews (with their given skills set) encounter problems meeting optimal post-ROSC targets in patients suffering from OHCA, and to investigate if this can be predicted based on patient-, provider- or treatment factors.

Study design: Prospective cohort study of all patients attended by the EMS services with an OHCA who regain ROSC and are transported to a single university hospital, in order to identify those patients with a ROSC after a non-traumatic OHCA who had deranged physiology and/or complications from OHCA EMS personnel was unable to prevent/deal with in the prehospital environment.

Study population: Patients, >18 years, transported by the EMS services to the ED of the University Hospital Groningen (UMCG) with a ROSC after OHCA in a 1 year period

Main study parameters/endpoints: Primary endpoint of our study is the percentage of OHCA patients with a prehospital ROSC who arrive in hospital with either a deranged physiology or with complications from OHCA EMS personnel was unable to deal with.

ELIGIBILITY:
Inclusion criteria:

* Non-traumatic OHCA (as confirmed in notes of ambulance crew) with ROSC obtained before transport to hospital
* Age > 18

Exclusion criteria:

* Traumatic cause of arrest (NB asphyxia due to hanging, electrocutions and drowning are not considered as traumatic arrests in this study, as normal ALS algorithms (special circumstances) are followed for these patients
* No ROSC before leaving OHCA
* Age <18
* Informed opt out of medical research of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years) patients with ROSC after OHCA transported to University Hospital Groningen by the EMS services.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
percentage of OHCA patients with a prehospital ROSC who arrive in hospital with either a deranged physiology or with complications from OHCA EMS personnel was unable to deal with | From pre-hospital ROSC to arrival at ED, approximately 1-2 hours
  Any of the below 5 minutes or more after ROSC is obtained:
  * -Airway intervention (SGA or ETT) not performed (when deemed necessary)
  * Actively Vomiting in absence of ETT after ROSC B: -Hypoxia: -SaO2 <94% on at least two consecutive readings
  * Hypercarbia: -ETCO2>5.5 kPa on at least two consecutive readings** C: -Low cardiac output: -Re-arrest during transport to hospital
  * ETCO2<3.0 on two consecutive readings
  * MAP<65mmHg on two consecutive readings
  * SBP<100 mmHg on two consecutive readings upon arrival in ED D: -Hypoxic agitation upon arrival in ED or uncontrolled prehospital hypoxic agitation despite benzodiazepine administration or when benzodiazepines contraindicated)
  * Seizures during transport E: -Hyperthermia

SECONDARY OUTCOMES:
Duration of period with deranged physiology, measured from moment of first occurrence until resolved or until arrival in hospital. | From pre-hospital ROSC to arrival at ED, approximately 1-2 hours
  Any of the following measured in minutes:
  * -Airway intervention (SGA or ETT) not performed (when deemed necessary)
  * Actively Vomiting in absence of ETT after ROSC B: -Hypoxia: -SaO2 <94% on at least two consecutive readings
  * Hypercarbia: -ETCO2>5.5 kPa on at least two consecutive readings** C: -Low cardiac output: -Re-arrest during transport to hospital
  * ETCO2<3.0 on two consecutive readings
  * MAP<65mmHg on two consecutive readings
  * SBP<100 mmHg on two consecutive readings upon arrival in ED D: -Hypoxic agitation upon arrival in ED or uncontrolled prehospital hypoxic agitation despite benzodiazepine administration or when benzodiazepines contraindicated)
  * Seizures during transport E: -Hyperthermia
Patient- and resuscitation factors related to deranged physiology and/or complications in the post arrest phase | From pre-hospital ROSC to arrival at ED, approximately 1-2 hours
Opinion of EMS providers weather or not they felt they were able to provide optimal post arrest care | From pre-hospital ROSC to arrival at emergency department, approximately 1-2 hours
  Measured by a survey, filled out by EMS crew at arrival at ED
Comparison of primary outcome of secondary outcomes between post ROSC patients attended by EMS only vs EMS and HEMS | From pre-hospital ROSC to arrival at emergency department, approximately 1-2 hours
Frequency distribution of airway interventions (SGA or ETT) not performed (when deemed necessary) | From pre-hospital ROSC to arrival at emergency department, approximately 1-2 hours
  -Airway intervention (SGA or ETT) not performed (when deemed necessary) in ED. NB NOT change of SGA for ETT when SGA is functioning well
Frequency distribution of actively vomiting in absence of ETT after ROSC in prehospital setting | From pre-hospital ROSC to arrival at ED, approximately 1 to 2 hours
Frequency distribution of the presence of hypoxia | From pre-hospital ROSC to arrival at ED, approximately 1 to 2 hours
  SaO2 <94% on at least two consecutive readings
Frequency distribution of low cardiac output | From pre-hospital ROSC to ICU (or CCU) admission, up to about 1 hours
  Presence of one of the following:
  * Re-arrest during transport to hospital
  * ETCO2<3.0 on two consecutive readings
  * MAP<65mmHg on two consecutive readings 12
  * SBP<100 mmHg on two consecutive readings
Frequency distribution of hypoxic agitation upon arrival in ED or uncontrolled prehospital hypoxic agitation despite benzodiazepine administration or when benzodiazepines contraindicated) | From pre-hospital ROSC to arrival at ED, approximately 1-2 hours
  Assessed by physician who enrolls patient
Frequency distribution of seizures during transport | From pre-hospital ROSC to arrival at ED, approximately 1-2 hours
Frequency distribution of the presence of hyperthermia | From pre-hospital ROSC to arrival at ED, approximately 1-2 hours
  Defined as a temperature >37.5 celsius

CONTACTS AND LOCATIONS:
Overall Officials: Ewoud ter Avest, dr, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided